CLINICAL TRIAL: NCT03840356
Title: Comparison of Postoperative Pain Scores Reported by Patients to the Surgical Teams and Nursing Staff
Brief Title: Postoperative Pain Reported to Nurses and Physicians
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Benjamin K. Wilke, Assistant Professor of Orthopedics, Mayo Clinic
Other Study IDs: 18-004244
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Pain; Pain Control; Postoperative Pain
MeSH Terms: conditions — Pain; Agnosia; Pain, Postoperative | interventions — Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postoperative: The study will evaluate orthopedic postoperative patients during the hospitalization.
  Interventions: Other: Postoperative

INTERVENTIONS:
Other: Postoperative — No intervention is planned in the study. This study is simply evaluating the consistency with which patients report their pain levels to different members of the medical team.

SUMMARY:
Effective pain control following surgical procedures is a goal for both the patient as well as the medical staff caring for them. There have been numerous studies evaluating differing treatment pathways, but most studies have relied on the Visual Analog Scale (VAS) or Numerical Rating Scale (NRS) to evaluate outcomes. These scales are subjective score given by the patient with no objective data input, therefore making comparisons subject to possible bias. There are no known studies comparing the pain scores provided by the patient to the surgical team compared to the nursing staff caring for the patient. The aim will be to compare these values to see if patients are consistent in their pain rating.

DETAILED DESCRIPTION:
The project will be conducted as a prospective study comparing numerical rating scale pain scores reported by the patients to the surgical team and the nursing staff. All orthopedic inpatients will be eligible for the study. Subjects will not be consented for the study prior to data collection in order to prevent bias. At the conclusion of the patient's involvement in the study they will be informed that their data has been collected and will have the opportunity to opt out of the study, at which time the collected data will be destroyed.

Postoperatively the surgical team will ask the patient to provide a pain score during morning rounds as part of routine care. The pain score will be recorded by a member of the surgical team. Within 60 minutes of their rounds and prior to any pain inducing events (such as physical therapy or repositioning), the surgical team will ask the nurse caring for the patient to enter the room by his/her self and ask the patient the same routine questions including the pain score. The nurse will record the pain score. No member of the surgical team will enter the room while the nurse is present in order to prevent bias. This process will be repeated once a day up to three days for each patient after the patient's operation.

ELIGIBILITY:
Inclusion Criteria:

* All inpatient postoperative orthopedic patients will be eligible for the study.

Exclusion Criteria:

* If a patient is unwilling to participate in the study.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include all postoperative orthopedic patients during the hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pain score | 3 days
  Pain scores will be compared between those reported by the patient to the nurse and physician to evaluate for consistency. The visual analog scale (VAS) ranges from a minimum score of 0 representing "no pain at all" and a maximum score of 10 which represents "worst pain imaginable". The VAS is represented as a 100 mm horizontal line in increments of 10mm. Subjects indicate their pain level on the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Wilke, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided